CLINICAL TRIAL: NCT05108129
Title: Ultrasound-guided Modified Thoracoabdominal Nerves Block Through Perichondrial Approach(M-TAPA)Versus Oblique Subcostal Transversus Abdominis Plane Block(OSTAP) for Postoperative Analgesia of Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: USG-guided M-TAPA vs OSTAP Block in Patients Undergoing Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-2021/02
Record Dates: First submitted 2021-10-20; First posted 2021-11-04 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2021-10

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: modified-thoracoabdominal nerves block; oblique subcostal transversus abdominis plane block; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Allocation: Randomized Intervention Model: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blocks will be administered after induction of general Anesthesia so participants will be blinded to which intervention they have had.
  Study investigators will not be aware of what group the participant belongs to when assessing the patient at post-operative period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M-TAPA (Active Comparator): In the operating room, all of the patients will receive standard monitoring. An anesthesiologist will perform anesthesia inductions. After tracheal intubation, a linear probe will be placed in the sagittal direction at the 10th costal margin, and transversus abdominis, internal oblique, and external oblique muscles will be identified. A block needle will be inserted with in-plane technique and 25 ml 0.25% bupivacaine will be injected between the transversus abdominis muscle and the lower aspect of the costal cartilage. The same procedure will be repeated on the contralateral side. The pain intensity during rest and motion will be evaluated with the 0-10 Numeric Rating Scale (NRS). Patients will receive standard multimodal analgesia comprising paracetamol, dexketoprofen, and tramadol.
  Interventions: Procedure: M-TAPA block
- Group OSTAP (Experimental): In the second group, the patients will receive oblique subcostal TAP block in the supine position immediately after the endotracheal intubation. The anesthesiologist of the operating room will place the ultrasound with a linear probe subcostally and from the xiphoid to the right iliac crest obliquely. Rectus abdominis muscle and underlying transversus abdominis muscle, will be identified near the costal margin. The needle will be directed to the transversus abdominis fascia. Local anesthetic solution of 25 ml 0.25% will be injected to between rectus abdominis and transversus abdominis muscles along the oblique subcostal line. The same procedure will repeated to the contralateral side. The pain intensity during rest and motion will be evaluated with the 0-10 Numeric Rating Scale (NRS). Patients will receive standard multimodal analgesia comprising paracetamol, dexketoprofen, and tramadol.
  Interventions: Procedure: OSTAP block

INTERVENTIONS:
Procedure: M-TAPA block — After tracheal intubation, a high-frequency linear probe will be placed in the sagittal direction at the 10th costal margin, and transversus abdominis, internal oblique, and external oblique muscles will be identified. A block needle will be inserted with in-plane technique and 25 ml 0.25% bupivacaine will be injected between the transversus abdominis muscle and the lower aspect of the costal cartilage. The same procedure will be repeated on the contralateral side.
  Standard perioperative and postoperative multimodal analgesia The pain intensity during rest and motion will be evaluated with the 0-10 Numeric Rating Scale (NRS). Patients will receive standard multimodal analgesia comprising paracetamol, dexketoprofen, and tramadol.
  Other Names: Global Quality of Recovery-15 score; Standard Pain Follow up and Monitorization
  Arms: Group M-TAPA
Procedure: OSTAP block — The patients will receive oblique subcostal TAP block in the supine position immediately after the endotracheal intubation. The anesthesiologist of the operating room will place the ultrasound with a linear probe subcostally and from the xiphoid to the right iliac crest obliquely. Rectus abdominis muscle and underlying transversus abdominis muscle, will be identified near the costal margin. The needle will be directed to the transversus abdominis fascia. Local anesthetic solution of 25 ml 0.25% will be injected to between rectus abdominis and transversus abdominis muscles along the oblique subcostal line. The same procedure will repeated to the contralateral side.
  Standard perioperative and postoperative multimodal analgesia The pain intensity during rest and motion will be evaluated with the 0-10 Numeric Rating Scale (NRS). Patients will receive standard multimodal analgesia comprising paracetamol, dexketoprofen, and tramadol.
  Other Names: Global Quality of Recovery-15 score; Standard Pain Follow up and Monitorization
  Arms: Group OSTAP

SUMMARY:
In this study, the postoperative analgesic effect of ultrasound-guided modified thoracoabdominal nerves blocks through perichondrial approach (M-TAPA) and oblique subcostal transversus abdominis plane block(OSTAP) will be searched in patients recruiting for laparoscopic cholecystectomy (LC) and the two groups will be compared in terms postoperative opioid consumption.

The primary aim of this study is to compare the effects of ultrasound-guided (M-TAPA) and OSTAP blocks on opioid consumption after LC surgery. It is hypothesized that M-TAPA will reduce opioid consumption of the patients more than the OSTAP block.

DETAILED DESCRIPTION:
Laparoscopy is a minimally invasive procedure, but postoperative pain is still the most common symptom after laparoscopic cholecystectomy (LC).

Oblique subcostal transversus abdominis plane (OSTAP) block is a regional anesthesia technique defined for abdominal surgeries. Previously, several studies have reported that ultrasound-guided OSTAP blocks reduce postoperative pain scores after LC. M-TAPA block is performed by applying local anesthetic to the lower surface of the chondrium. This technique provides effective analgesia in the abdominal wall.

This study will be conducted as a single-center, prospective, randomized, double-blinded trial in a university hospital. Patients scheduled for elective laparoscopic cholecystectomy will be screened for enrollment in the study. After randomization, M-TAPA and OSTAP blocks will be performed under ultrasound guidance after administering general anesthesia and prior to the skin incision. An anesthesiologist who performed blocks will not involve in the data collection. Other health care workers who will involve in the evaluation of postoperative pain scores, vital parameters, nausea and vomiting, antiemetic, opioid consumption, and Quality of Recovery score will be blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age between 18 and 70 years with American Society of Anesthesiology (ASA) physical status I-II, who will be scheduled for an elective laparoscopic cholecystectomy surgery included in the study

Exclusion Criteria:

* presence of coagulation disorder
* infection at the injection site of the block
* known allergy to local anesthetics
* advanced hepatic or renal failure
* can not communicate in Turkish
* history of abdominal surgery or trauma
* conversion of laparoscopic to open surgery
* consumption of any pain killers within the 24 h before the operation
* chronic opioid consumption
* pregnancy
* alcohol or drug abuse
* body mass index (BMI) ≥ 35 kg m-2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Total daily consumption of rescue analgesic | Postoperative 24 hours
  If Numerical Rating Scale (NRS) score of the patient is equal to or over 4, IV 50 mg tramadol will be applied as a rescue analgesic.

SECONDARY OUTCOMES:
Numerical Rating Scale scores | Postoperative 24 hours
  Numerical Rating Scale scores will be evaluated both at rest and motion. A blinded anesthesiologist will assess postoperative pain during rest and motion at the postoperative 15th,30th and 60th minute, second, 6th, 12th, and 24th hour by using an 11-point Numerical Rating Scale which ranges from '0' (means no pain) to '10' (means worst pain imaginable).
Time to first rescue analgesic | Postoperative 24 hours
  The time for administration of first rescue analgesic.
Adverse events | Postoperative 24 hour
  Incidence of nausea and vomiting during postoperative 24 hour time period will be noted.
Metoclopromide consumption | Postoperative 24 hour
  The severity of the nausea will be assessed on a 4 -point scale (0=none 1=mild, 2=moderate 3=severe). If the patients nausea score is ≥2 the patient will receive 10 mg metoclopromide.
Sedation score | Postoperative 24 hour
  Sedation level of the patients will be assessed on a 4-point scale (0=alert, 1=sleepy, easy to arouse verbally, 2= drowsy, 3=does not open eyes to verbal commands) at postoperative 15th,30th and 60th minute, second, 6th, 12th and 24th hour.
Quality of recovery levels between groups by using QoR-15 questionnaire | Postoperative 24th hour
  A 15-parameter Quality of Recovery score (QoR-15) has been recommended as the optimum tool to evaluate overall patient-centers measures of recovery after surgery, including pain. It is a questionnaire that is given to patients to do postoperatively and is scored from 0 to 150 where 150 indicates that the patient has had an excellent recovery QoR-15 score will be recorded on the morning of operation and at the postoperative 24th hour.
Anesthetized thoracoabdominal areas at 2 hours after surgery | Postoperative 2 hours
  The blinded anesthesiologist will assess sensory levels using pinprick test postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Basaran, MD,DESA, Study Director — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

REFERENCES:
- [Derived] Bilge A, Basaran B, Altiparmak B, Et T, Korkusuz M, Yarimoglu R. Comparing ultrasound-guided modified thoracoabdominal nerves block through perichondrial approach with oblique subcostal transversus abdominis plane block for patients undergoing laparoscopic cholecystectomy: a randomized, controlled trial. BMC Anesthesiol. 2023 Apr 27;23(1):139. doi: 10.1186/s12871-023-02106-z. PMID 37106319